CLINICAL TRIAL: NCT00236717
Title: TOPAMAX (Topiramate) Monotherapy Comparison Trial to Standard Monotherapy in the Treatment of Newly Diagnosed Epilepsy (RWJ-17021-000); Phase IIIB
Brief Title: A Study of the Effectiveness and Safety of Topiramate Compared With a Standard Therapy in Patients Newly Diagnosed With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005461
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Seizures
Keywords: Epilepsy; Seizures; Topiramate; Prophylaxis; Antiepileptic
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Topiramate; Carbamazepine; Valproic Acid

INTERVENTIONS:
Drug: Topiramate; Carbamazepine; Valproate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of topiramate to standard antiepileptic drugs in children and adults with newly diagnosed epilepsy.

DETAILED DESCRIPTION:
Topiramate is a drug that is currently widely used for the treatment of seizures in adults and pediatric patients (2 to 16 years of age). This is a randomized, double-blind, parallel-group study to evaluate the effectiveness and safety of two dosages of topiramate (100 or 200mg per day) compared with standard antiepileptic drugs (carbamazepine or valproate) in patients with newly diagnosed epilepsy. The study is composed of three phases: baseline (up to 7 days), double-blind treatment, and a blinded extension. The double-blind phase is divided into two periods: titration, in which the dose of drug is gradually increased (approximately 35 days), and stabilization (of variable duration, with regular scheduled visits up to 92 days and then every 3 months thereafter). The dose of study drug remains constant during the stabilization period. In the blinded extension, patients completing the double blind phase are given the opportunity to take the other study medication in a blinded fashion (patient unaware of identity of the drug). This phase continues until the patient leaves the study or the data base for the double blind phase is finalized. The primary assessment of effectiveness is the time to first seizure from Day 15 of the study. Safety assessments include the frequency of adverse events during the study, results of clinical laboratory tests (hematology and biochemistry), measurements of vital signs and body weight, and physical examination findings. The study hypothesis is that the 200mg dose of topiramate is superior to the 100mg dose in delaying the time to first seizure and is well-tolerated. Oral topiramate (25milligram [mg] or 50mg capsules or tablets),starting at 25mg/day (Week 1),increasing to 100mg or 200mg/day (Week 5).Increasing carbamazepine to 600mg/day or valproate to 1250mg/day (Week 5).Maximum dosages continue for a variable time and then taper over 4 weeks to starting dose.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 30 kilograms
* New epilepsy diagnosis and at least one unprovoked seizure within 3 months before study entry
* No history of antiepileptic drug use or taking a single antiepileptic drug for no longer than 6 weeks
* Females must be sexually abstinent, surgically sterile, or using adequate birth control measures, and have a negative pregnancy test before study entry

Exclusion Criteria:

* Patients who do not have epilepsy
* Have progressive or degenerative disorders (for example, certain hereditary conditions)
* Have a significant history (within last 2 years) of unstable medical diseases (heart, kidney, hormone, or liver diseases)
* Have mental retardation or other condition that could make interpretation of the study results difficult
* alcohol or drug abuse within the previous year

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 1997-09; Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Time to first seizure from Day 15 of the study

SECONDARY OUTCOMES:
Time to first seizure from Day 1 of the study; time to exit from the study; proportion of seizure-free patients during the last 6 months of the double-blind period; safety evaluations conducted throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Wheless JW, Neto W, Wang S; EPMN-105 Study Group. Topiramate, carbamazepine, and valproate monotherapy: double-blind comparison in children with newly diagnosed epilepsy. J Child Neurol. 2004 Feb;19(2):135-41. doi: 10.1177/08830738040190020901. PMID 15072107
- See also: A study of the effectiveness and safety of topiramate compared with a standard single medicine therapy in patients newly diagnosed with epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=646&filename=CR005461_CSR.pdf